CLINICAL TRIAL: NCT06290609
Title: Control of Incomplete Spinal Cord Injury-Related Spasticity by Means of Vibrotactile Coordinated Reset Fingertip Stimulation
Brief Title: Vibrotactile Coordinated Reset for Spasticity After Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter Tass, MD, PhD, Protocol Director, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 72799
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-08

CONDITIONS: Spasticity, Muscle; Spinal Cord Injuries
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: A single group of participants who will receive active treatment with the experimental stimulation device will be studied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Vibrotactile Coordinated Reset stimulation (Experimental): Participants will receive vCR stimulation, involving vibratory stimulation of the fingertips, with the Stanford CR Glove on a daily or weekly basis.
  Interventions: Device: Vibrotactile Coordinated Reset

INTERVENTIONS:
Device: Vibrotactile Coordinated Reset — The experimental device, the Stanford CR Glove, is designed to deliver vibratory stimulation to the fingertips of each hand according to a specific pattern, known as vibrotactile Coordinated Reset, which theoretically disrupts abnormal neuronal synchrony and is expected to restore function.

SUMMARY:
The purpose of our study is to evaluate vibrotactile Coordinated Reset (vCR) and its effects on spasticity symptoms in incomplete spinal cord injured patients. vCR will be administered with a device called the Stanford CR Glove. vCR is expected to provide patients with a non-invasive alternative to the most widely used treatments such as oral baclofen and or deep brain stimulation. Patients will be followed for three months and will be asked to come to the lab for clinical testing 4 times during this period. A total of 30 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment: Any adult ages 18 and over
2. Spinal Cord Injury: ASIA C or D injury at level C1-T1
3. Duration of incomplete spinal cord injury minimum 1 years clinical/fundamental
4. Spasticity with a of MAS score >3 present in upper extremities.
5. Fluent in English
6. If patient is on medication that affects brain function or alters EEG activity, the patient must feel comfortable going off this medication prior to EEG recording.
7. Appropriate social support if required during an off-medication state.
8. Comfortable with technology; can use a computer, check email, and access the internet; can initiate and engage in a virtual meeting for training and monitoring purposes.
9. Feels comfortable going off certain spasticity related medication during in-person study visits
10. Lives in the United States

Exclusion Criteria:

1. Sensory deficits in palma manus resulting in missing inter digit discrimination of the fingertips.
2. Any significant neuro-psychiatric problems, including acute confusional state, ongoing psychosis, or suicidal tendencies.
3. Any current drug or alcohol abuse.
4. Participation in another drug, device, or biologics trial concurrently or within the preceding 30 days. Any other trial participation should be approved by the Principal Investigators.
5. Pregnancy, breast-feeding or wanting to become pregnant.
6. Physical limitations unrelated to spasticity that would affect motor ratings.
7. Craniotomy
8. Brain surgery
9. Patient is unable to communicate properly with staff (i.e., severe speech problems)
10. Medications that may affect relevant synaptic plasticity
11. Concurrent Botox treatment
12. A type of hairstyle that would impede the use of an EEG cap.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in spasticity with the Modified Ashworth Scale (MAS) at 2 hours, 1 week, 4 weeks, and 12 weeks. | Baseline, 2 hours, 1 week, 4 weeks, and 12 weeks
  The MAS is a method of grading muscle spasticity according to a 6-point ordinal scale. In this assessment, spasticity is judged to be present when resistance is encountered during passive muscle stretching. With a score of 0 indicating no increase in muscle flexion and a score on 4 indicating and increase in muscle flexion. Low numeric ratings indicate better outcomes and high numbers indicate worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided